CLINICAL TRIAL: NCT00971373
Title: Pilot Study to Determine the Effectiveness of Antimicrobial Scrubs on Bacterial Burden of HCW's Hands and Clothing in a Clinical Setting
Brief Title: Pilot Study to Determine the Effectiveness of Antimicrobial Healthcare Worker's (HCW) Hands and Clothing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HM12358
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Effectiveness of Antimicrobial Impregnated Scrubs in a Healthcare Setting
Keywords: antimicrobial; epidemiology; bacteriology; CFU
MeSH Terms: interventions — Nanospheres

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exp Scrubs (Experimental): antimicrobial impregnated scrubs
  Interventions: Other: Vestagen scrubs
- Non-antimicrobial scrubs (No Intervention): Non-antimicrobial scrubs

INTERVENTIONS:
Other: Vestagen scrubs — antimicrobial impregnated textile
  Other Names: Vestagen; Nanosphere
  Arms: Exp Scrubs

SUMMARY:
This is a pilot study to determine the effectiveness of antimicrobial scrubs on bacterial burden of HCW's hands and clothing in a clinical setting.

DETAILED DESCRIPTION:
Goals of the pilot study:

* Compare CFU counts on antimicrobial vs standard scrubs in a clinical setting
* Assess CFU counts on the hands of HCWs wearing antimicrobial vs non-antimicrobial scrubs
* Assess HCW hand hygiene compliance during the study protocol
* Correlate device associated infection rates during protocol to historical controls
* Assess feasibility of applying protocol to a longer,12-24 month, prospective crossover-trial to definitively study and assess the impact of antimicrobial scrubs on HCW apparel and hand colonization, control of multi-drug resistance organisms, hand hygiene compliance, and device associated hospital acquired infection rates.

II. Design

Cross-over trial in an ICU or Hospital Ward

III. Outcome Measures

1. CFU count on participants

   1. Hands
   2. Scrubs
   3. Antimicrobial scrubs vs standard scrubs
2. Hand Hygiene Compliance
3. Device associated nosocomial infections rates

ELIGIBILITY:
Inclusion Criteria:

* HCWs in the MRICU

Exclusion Criteria:

* Under the age of 18 who is not a healthcare worker in the MRICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Antimicrobial impregnated scrubs | 4 months

SECONDARY OUTCOMES:
HCW hand and scrub average bacterial counts | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Bearman, M.D., MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States